CLINICAL TRIAL: NCT05438355
Title: The Effect of Polycystic Ovary Syndrome on the Morphokinetics or Abnormalities on Early Embryonic Development: a Time Lapse Study
Brief Title: The Effect of Polycystic Ovary Syndrome on the Embryo Morphokinetics ( PCOS )
Status: Completed | Type: Observational
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2022JIAI-06
Record Dates: First submitted 2022-06-21; First posted 2022-06-29 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: PCOS
Keywords: PCOS; Time-lapse; Infertility; Morphokinetics
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The infertility women with PCOS: Infertile women undergoing assisted reproduction were consecutively recruited at Ji Ai G-IVF institute from March 2021 to December 2021. Women aged < 38 years without endometriosis and more than 6 oocytes were retrieved . Patients were divided in PCOS according to the Rotterdam criteria for PCOS, defined by the presence of anovulation and polycystic ovaries.
- The infertility women without PCOS: Infertility women with fallopian tubal factor infertility and with normal menstrual cycles were undergoing IVF/ICSI cycles at Shanghai Ji Ai G-IVF institute from March 2021 to December 2021.Women aged < 38 years without endometriosis and more than 6 oocytes were retrieved.

SUMMARY:
Polycystic ovarian syndrome (PCOS) is a complex endocrine and metabolic syndrome which accounts for 75% of women with anovulatory infertility. The cause of infertility in PCOS is already unknown. Although efforts have been made, many PCOS patients turned out to have worse oocyte maturity and IVF outcomes. Time-lapse analysis of embryo development can detect the abnormal timeline and cleavage mode which may affect the embryo viability of PCOS. However, there are still some debates on the effect of PCOS on the early embryo development by time-lapse analysis.

DETAILED DESCRIPTION:
Method:

A consecutive cohort of 153 infertile women attending In vitro fertilization (IVF) or Intra-cytoplasmic sperm injection (ICSI) treatment at Shanghai Ji Ai G-IVF institute was requited from March 2021 to December 2021. During the period, couples undergoing IVF/ICSI treatment were offered blastocyst culture to day 6 and time-lapse imaging (TLI) as part of a study evaluating parameters for embryo selection. Women aged < 38 years without endometriosis and with more than 6 oocytes retrieved were eligible. Patients were categorized in two groups. Women with regular menstrual cycles and no clinical signs of PCOS (non-PCOS) and women fulfilling the Rotterdam diagnostic criteria for PCOS detected by the presence of anovulation and polycystic ovaries (PCO), which was diagnosed by luteal-phase progesterone testing and trans-vaginal ultrasound, respectively. Biochemical parameters of androgen excess were included in the diagnosis when available, whereas subjective symptoms of androgen excess (acne, hirsutism, alopecia) were not included. Ethical approval Written informed consent was obtained from all patients before inclusion. Shanghai Ji Ai ethical Committees approved the study.

Ovarian stimulation:

Patients were treated with individual doses of gonadotropin, based on serum anti-mullerian hormone (AMH) and/or antral follicle count. Patients were stimulated by gonadotropin-releasing hormone (GnRH) antagonist protocol using rec-follicle stimulating hormone (FSH) or human menopausal gonadotropin (HMG) for stimulation according to clinical guidelines. A dose of 10,000 IU of human chorionic gonadotropin (hCG) was administered when at least 3 follicles measured ≥ 17 mm, and ultrasound guided oocyte retrieval was conducted 36 h later. Oocyte retrieval and ICSI/IVF Ovarian stimulation and oocyte retrieval were performed according to standard procedures. After fertilization, ICSI embryos were immediately placed in the time-lapse incubator (EmbryoScope™). IVF embryos were cultured for approximately 18 h in a conventional incubator. Before IVF embryos were transferred to the EmbryoScope, adhering cumulus cells were removed to ensure optimal image acquisition. In the EmbryoScope, all embryos were cultured until arrest or removal at day 6.

Embryo assessment:

All embryos with 2 pronuclei completing the first cleavage were annotated manually. The following parameters were annotated with time points: appearance and disappearance of 1st nucleus and 2nd nucleus after 1st division, 1st - third divisions and blastocyst. All time-points were normalized to first cleavage and treated as durations for further analysis in order to overcome the limitation of inexact starting points, and facilitate comparison between IVF and ICSI populations. For the same reason, no parameters before first cleavage were investigated. Durations of cell cycles and cell stages were subsequently calculated as the interval between two time-points. Two parameters (multi-nucleation and direct cleavage to 3-cell stage) were assessed by binary values yes and no. Embryos were selected for transfer according to conventional measures of morphological quality on day 6 according to the Gardner criteria. No time-lapse parameters were used in the selection process. The observer was blinded to the patient's treatment data and medical history.

Statistics:

The influence of PCOS on embryo development was tested in regression models for clustered data. A covariance regression model was used to account for potential confounding variables: female age, BMI and fertility treatment. In total, 768 embryos from 80 PCOS women, and 676 embryos from 73 non-PCOS women were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women aged < 38 years without endometriosis and with more than 6 oocytes retrieved were eligible.

Exclusion Criteria:

* All embryos with more or less than 2 pronuclei, and that did not undergo first cleavage were excluded

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertility patients udergoing IVF/ICSI cycles at Shanghai JiAi G-IVF institute from March 2021 to December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Embryonic developmental timing | From fertilization until transfer at day 6
  Embryonic developmental timing assessed by Time-lapse analysis

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Sun, PHD, Study Chair — Shanghai G-IVF institute
Locations (1):
- Ji Ai Genetics and IVF center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Result] Kirkegaard K, Kesmodel US, Hindkjaer JJ, Ingerslev HJ. Time-lapse parameters as predictors of blastocyst development and pregnancy outcome in embryos from good prognosis patients: a prospective cohort study. Hum Reprod. 2013 Oct;28(10):2643-51. doi: 10.1093/humrep/det300. Epub 2013 Jul 30. PMID 23900207
- [Result] Gardner DK, Surrey E, Minjarez D, Leitz A, Stevens J, Schoolcraft WB. Single blastocyst transfer: a prospective randomized trial. Fertil Steril. 2004 Mar;81(3):551-5. doi: 10.1016/j.fertnstert.2003.07.023. PMID 15037401